CLINICAL TRIAL: NCT06140017
Title: Achieving Sustained Early Child Development Impacts at Scale: A Test in Kenya
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Early Childhood Development Network for Kenya (ECDNeK) (Unknown); Safe Water and AIDS Project (Other)
Responsible Party: Principal Investigator, Italo Lopez Garcia, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD107116 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Child Development; Child Behavior; Language, Child
MeSH Terms: conditions — Child Behavior; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- In-Person Group Delivery (Active Comparator): A total of 30 villages will receive a traditional in-person group-based delivery for Msingi Bora, an ECD parenting intervention featuring 16 biweekly village sessions over 8 months, followed by monthly "booster" meetings for 16 additional months. Sessions will be delivered within by existing village Community Health Volunteers (CHVs). Mothers and children will be invited to attend a total of 32 in-person sessions of roughly 1.5-2 hours apiece over 24 months.
  Interventions: Behavioral: Msingi Bora responsive parenting and family wellbeing program
- Hybrid mHealth/In-Person Group Delivery (Experimental): 30 CHVs will deliver a hybrid intervention that combines in-person meetings with remote delivery for Msingi Bora, an ECD parenting intervention. Mother-child dyads will be invited to participate in roughly 10 in-person group sessions in the first 8 months, followed by 5 in-person group sessions over the next 16 months. For those sessions delivered remotely, mothers will receive videos demonstrating the practices, SMS messages, be invited to participate in group SMS/WhatsApp chats with the CHV and other village mothers, and periodic phone calls. The project will provide smartphones to all mothers assigned to this arm for facilitation.
  Interventions: Behavioral: Msingi Bora responsive parenting and family wellbeing program
- Control Group (No Intervention): Mothers and children in 30 villages will not receive any intervention beyond information about child feeding during a baseline survey.

INTERVENTIONS:
Behavioral: Msingi Bora responsive parenting and family wellbeing program — Msingi Bora's structured curriculum of 16 biweekly sessions and monthly boosters thereafter are organized around five key messages: love and respect within the family, responsive talk, responsive play, hygiene, and nutrition.
  Arms: Hybrid mHealth/In-Person Group Delivery; In-Person Group Delivery

SUMMARY:
An estimated 43% of children under age 5 in low- and middle-income countries (LMICs) experience compromised development due to poverty, poor nutrition, and inadequate psychosocial stimulation. Numerous early childhood development (ECD) parenting interventions have been shown to be effective at improving ECD outcomes, at least in the short-term, but they are a) still too expensive to implement at scale in low-resource and rural settings, and b) their early impacts tend to fade over time in the absence of continued support. New ways to deliver effective ECD parenting interventions are sorely needed that are both low-cost to be potentially scalable, while also able to sustain impacts long-term.

The rapid growth and low cost of mobile communications in LMIC settings presents a potentially promising solution to the competing problems of scalability and sustainability. Yet there is no rigorous research on mobile-health (mHealth) interventions for ECD outcomes in LMIC settings. Study investigators recently showed that an 8-month ECD parenting intervention featuring fortnightly group meetings delivered by Community Health Workers (CHWs) from Kenya's rural health care system significantly improved child cognitive, language, and socioemotional development as well as parenting practices, and a group-based delivery model was more cost-effective than previous ECD interventions. Yet it is still too expensive for scaling in a rural LMIC setting such as rural Kenya, particularly if interventions are needed that can be extended for longer periods of time to increase their ability to sustain impacts. This study will experimentally test a traditional in-person group-based delivery model for an ECD parenting intervention against an mHealth-based delivery model that partially substitutes remote delivery for in-person group meetings. The relative effectiveness and costs of this hybrid-delivery model will be assessed against a purely in-person group model, and the interventions will extend over two years to increase their ability to sustain changes in child outcomes longer-term. The evaluation design is a clustered Randomized Control Trial across 90 CHWs and their associated villages and 1200 households. The central hypothesis is that a hybrid ECD intervention will be lower cost, but remote delivery may be an inferior substitute for in-person visits, leaving open the question of the most cost-effective program.

ELIGIBILITY:
Inclusion Criteria:

* mothers or other primary caretakers aged 18 years or older
* able to read English or Swahili at a level sufficient to understand the SMS messages
* with a child aged 6-18 months at recruitment without signs of severe mental or physical impairments (youngest child if more than one eligible for a given mother)

Exclusion Criteria:

* mothers/households without children
* households with children that are outside the age range of 6-18 months at baseline
* mothers who lack basic literacy so as not to understand SMS messages

Min Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Child Cognitive Development - Bayley | Midline/8-month survey, Endline/24-month survey
  The Bayley Scales of Infant Development 3rd edition (Bayley's III) is validated in African settings and provides measures for all dimensions of child development up to 42 months of age. The official age-standardized cognitive scale has a 0-19 range with higher values denoting better scores.

SECONDARY OUTCOMES:
Parenting Behaviors | Midline/8-month survey, Endline/24-month survey
  The Home Observation for Measurement of the Environment (HOME)- Short Form (SF) inventory has four versions: one for children under age three; a second for children between the ages of three and five; a third for children ages six through nine; and a fourth version for children ten and over. The total raw score for the HOME-SF is a simple summation of the recorded individual item scores and it varies by age group, as the number of individual items varies according to the age of the child. At the endline/month 8 survey the HOME scale scores will range from 0-45, with higher scores denoting better outcomes.

OTHER OUTCOMES:
Maternal Depression | Midline/8-month survey, Endline/24-month survey
  The Patient Health Questionnaire (PHQ-8) is a self-reported measure of depressive symptoms during the previous two weeks. It is composed of 8 Likert-style items with a response scale ranging from 0 (Not at all) to 3 (Nearly every day). The PHQ-8 final score ranges from 0 to 24, with higher scores corresponding to higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Lopez Garcia, PhD, Principal Investigator — University of Southern California; Jill E Luoto, PhD, Principal Investigator — University of Southern California
Locations (1):
- Safe Water and AIDS Project, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be stripped of identifiers prior to release for sharing. In no way will there be the possibility of deductive disclosure of subjects. We will make the data without identifiers publicly available in accordance with NIH policy by posting it in de-identified form to the Inter-university Consortium for Political and Social Research (ICPSR) data bank. More information on their data confidentiality practices can be found at: https://www.icpsr.umich.edu/web/pages/datamanagement/confidentiality/index.html.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Garcia IL, Luoto J, Aboud F, Jervis P, Mwoma T, Alu E, Odhiambo A. In-person versus remote (mHealth) delivery for a responsive parenting intervention in rural Kenya: a cluster randomized controlled trial. BMC Public Health. 2024 Sep 5;24(1):2421. doi: 10.1186/s12889-024-19828-5. PMID 39237936
- [Derived] Garcia IL, Luoto J, Aboud F, Jervis P, Mwoma T, Alu E, Odhiambo A. In-person versus remote (mHealth) delivery for a responsive parenting intervention in rural Kenya: A cluster randomized controlled trial. Res Sq [Preprint]. 2024 Aug 16:rs.3.rs-4733054. doi: 10.21203/rs.3.rs-4733054/v1. PMID 39184097